CLINICAL TRIAL: NCT01477905
Title: Study of Proper Operation of the Syringe Pump Used in Priming of the Syringe
Brief Title: Impact of Priming the Infusion System on the Performance of Target-controlled Infusion of Remifentanil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-DEV-DEO-11-005
Record Dates: First submitted 2011-11-14; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Intravenous Drug Usage
Keywords: priming; remifentanil; target-controlled infusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remi50 no prime (Experimental): For using experimental target control infusion device (TCIs), targeting an effect-site concentration (Ceff) of 4.0 ng/ml, were randomly performed using 50 μg/ml (Remi50) of remifentanil, and without PRIMING,
  Interventions: Device: Remi50 with prime
- Remi20 no prmie (Experimental): For using experimental TCIs, targeting an effect-site concentration (Ceff) of 4.0 ng/ml, was 20 μg/ml (Remi20) of remifentanil, and without PRIMING
  Interventions: Device: Remi20 with prime

INTERVENTIONS:
Device: Remi50 with prime — for using experimental TCIs, targeting an effect-site concentration (Ceff) of 4.0 ng/ml, was performed using 50 μg/ml (Remi50) of remifentanil, with PRIMING
  Other Names: remi50 prime
  Arms: Remi50 no prime
Device: Remi20 with prime — For using experimental TCIs, targeting an effect-site concentration (Ceff) of 4.0 ng/ml, was 20 μg/ml (Remi20) of remifentanil, and with PRIMING
  Other Names: remi20 prime
  Arms: Remi20 no prmie

SUMMARY:
The investigators attempted to determine an adequate priming volume for our infusion system, and investigated the extent of a possible delay of the drug effect, that would result from mechanical defects of the infusion system, with or without priming the infusion system, using direct gravimetrical measurements of virtual infusate amounts during target controlled infusion of 2 remifentanil diluents.

DETAILED DESCRIPTION:
Priming the infusion system (PRIMING) was performed using an evacuation of 2.0 ml to the atmosphere prior to Target-controlled Infusion (TCI). Forty eight TCI, using 50 μg/ml or 20 μg/ml of remifentanil diluents, were performed targeting 4.0 ng/ml of effect site concentration (Ceff), with or without PRIMING. Using simulations, the gravimetrical measurements of the delivered infusates reproduced actual predicted concentrations.

ELIGIBILITY:
Inclusion Criteria:

* electric medical records of the patients who had undergone general anaesthesia

Exclusion Criteria:

* body weight exceeding 20% of ideal body weight

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
delivered infusates of remifentanil | base line from 30 min of TCI was maintained
  For targetting an effect-site concentration (Ceff) of 4.0 ng/ml, were randomly performed using 50 μg/ml (Remi50) or 20 μg/ml (Remi20) of remifentanil, and with or without PRIMING, TCI data files, including predicted plasma (Cp-proper), and effect-site (Ceff-proper) concentrations were saved

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, M.D., Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea

REFERENCES:
- [Result] Swinhoe CF, Peacock JE, Glen JB, Reilly CS. Evaluation of the predictive performance of a 'Diprifusor' TCI system. Anaesthesia. 1998 Apr;53 Suppl 1:61-7. doi: 10.1111/j.1365-2044.1998.53s104.x. PMID 9640119